CLINICAL TRIAL: NCT07326657
Title: Open-label, Controlled, Randomized, Multicenter Study Evaluating Intact Fish Skin Graft in Promoting AutoLOgous Skin Tissue ReGeneratIon of Deep Partial-Thickness Burns: The LOGI Study
Brief Title: Evaluating Whether Intact Fish Skin Graft Can Decrease the Need for Autograft in the Treatment of Deep Partial-Thickness Burns
Acronym: LOGI
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Kerecis Ltd. (Industry)
Collaborators: American Burn Association (Other); BData, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KS-1040
Record Dates: First submitted 2025-06-03; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Partial-thickness Burn Wounds
Keywords: burn; deep partial-thickness; Kerecis; fish skin graft; autograft; split thickness skin graft; fish skin
MeSH Terms: conditions — Burns; Ichthyosis Vulgaris | interventions — Transplantation, Autologous

STUDY DESIGN:
Intervention Model Description: The intervention study model is a split-body intervention in which each patient has part of their burn treated with intact fish skin graft and another part treated with autograft as the standard-of-care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- IFSG-Treated Area of Burn (Experimental): The area of the deep partial-thickness burn that is treated with IFSG
  Interventions: Device: Intact fish skin graft
- SOC Autograft-Treated Area of Burn (Active Comparator): The area of the deep partial-thickness burn that is treated with autograft as standard-of-care
  Interventions: Procedure: autograft

INTERVENTIONS:
Device: Intact fish skin graft — Treatment with IFSG
  Arms: IFSG-Treated Area of Burn
Procedure: autograft — Treatment with autograft
  Arms: SOC Autograft-Treated Area of Burn

SUMMARY:
The goal of this randomized controlled clinical trial is to determine whether use of Kericis Intact Fish Skin Graft (IFSG) can decrease the amount of autograft tissue needed for treatment of deep partial-thickness burns in patients at least 18 years of age with a deep partial-thickness burn for whom autograft treatment is clinically indicated. This clinical trial seeks to collect the following:

1. Difference in the percentage area of the IFSG treatment site and control autograft treatment site that required autografting within 1 month of treatment
2. Proportion of subjects achieving durable wound closure of the IFSG treatment site without autograft placement within 2 months of treatment
3. Difference in cosmesis between the IFSG treatment site and autograft treatment site a year after treatment
4. Difference in the pain intensity between the IFSG treatment site and autograft treatment site

Each participant will receive autograft and intact fish skin graft (IFSG) on different areas of their deep partial-thickness burn. Participants will be assessed for the need for further autograft treatment. Participants will also be assessed for wound closure, pain, and cosmesis.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at time of consent
2. Must have thermal burn(s) with intact dermal elements for which excision and autografting are clinically indicated.
3. Be able to provide written informed consent or have a legally authorized representative
4. Have sufficient healthy skin identified and designated as a potential donor site in the event that the IFSG treatment site requires autografting.
5. Investigator expects that the donor site will heal without grafting
6. Have a complex skin defect of 3 to 49% Total Body Surface Area, which can consist of more than one contiguous area

   At the time of debridement:
7. Have thermal burn(s) with intact dermal elements for which excision and autografting are clinically indicated
8. Study treatment areas can be up to 2000 cm2
9. Must have at least 100 cm2 TBSA for which autografting is indicated and on which IFSG can be applied, which may be composed of up to 3 non-contiguous areas located on the same extremity or plane of the torso
10. Application of IFSG or SOC must be initiated within 14 days of injury (Application of IFSG or SOC must be initiated within 14 days of injury)
11. Have first excision and grafting of study treatment sites
12. Have thermal burn(s) on the torso or extremities

Exclusion Criteria:

1. Known allergy or hypersensitivity to fish (shellfish allergy is OK)
2. Female who is actively pregnant or currently breast-feeding
3. Vulnerable populations
4. Currently receiving systemic immunosuppressive therapy
5. Current or known history of malignancy or receipt of chemotherapy
6. History of Diabetes with documented uncontrolled diabetes (as defined by an A1C >9) within the last 6 months
7. Have an expected survival of less than 3 months
8. Are currently participating/have participated in the treatment group of an interventional study within 90 calendar days prior to consent
9. Have other wounds present for > 30 days

   At the time of debridement:
10. Treatment area is assessed as full-thickness after debridement
11. Treatment areas on the face, neck, head, hands, feet, buttocks, perineum, and areas over joints (Treatment areas may only be on the torso or extremities)
12. Have a clinical or laboratory determination of infection at the anticipated treatment sites.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Difference in percentage area of the IFSG treatment site and control autograft treatment site that required autografting by 1 month. | From initial surgical IFSG/autograft treatment post-enrollment to 28 +/- 3 days later

SECONDARY OUTCOMES:
Proportion of subjects achieving durable wound closure of the intact fish skin treatment site at Month 2 without autograft placement | From initial treatment with IFSG/autograft post-enrollment to 60 +/- 7 days later
Difference in cosmesis between the IFSG treatment site and autograft treatment site at Month 12 based on observer POSAS total score | From initial treatment with IFSG/autograft post-enrollment to 365 +/- 30 days later
  Scar quality will be assessed using the Patient and Observer Scar Assessment Scale (POSAS) that describes scar quality on a scale from 1-10 with 1 being a scar very similar to normal skin and 10 being a severe scar very unlike normal skin.
Difference in the pain intensity between the IFSG treatment site and autograft treatment site one week after treatment based on the Wong-Baker FACES pain rating scale (FPRS) | From initial treatment with IFSG/autograft post-enrollment to 7 +/- 1 days later
  The Wong-Baker FACES pain rating scale presents a range of faces with a happy face associated with a score of 0, meaning "no hurt", to a very sad face associated with a score of 10, meaning "hurts worst."

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided